CLINICAL TRIAL: NCT00673998
Title: The Effects of Rest Interval on Quadriceps Torque During an Isokinetic Testing Protocol in Elderly and Young Men
Brief Title: Isokinetic Testing Protocol in Elderly and Young Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Brasilia (Other)
Responsible Party: Martim Bottaro, PhD, University of Brasilia
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UCB-072/2004
Record Dates: First submitted 2008-04-30; First posted 2008-05-07 (Estimated); Last update posted 2008-05-07 (Estimated); Status verified 2008-05

CONDITIONS: Healthy
Keywords: Isokinetic; Fatigue; Strength; Older
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Isokinetic Dynamometer (Biodex system III) — Biodex system III Isokinetic Dynamometer (Biodex Medical, Inc., Shirley, NY).
  Other Names: Biodex Isokinetic Dynamometer; Cybex Isokinetic Dynamometer

SUMMARY:
An age-related decrease in muscular strength may have a detrimental effect on muscle fatigue and recovery. To date, only one study has determined the effect of varied rest intervals (RI) between exercise sets in active younger and older women. They reported that active younger and older women require similar RI between sets to recovery full isokinetic knee extension peak torque (PT). However, we are unaware of any published studies comparing RI PT recovery between younger and older men. Thus, the purpose of this study was to compare the effect of two different RI's between sets of isokinetic knee extension exercise on PT, and Total Work (TW) between untrained younger and older men.

DETAILED DESCRIPTION:
18 young men (24.22 ± 2.58 yrs) and 20 older men (66.85 ± 4.02 yrs) performed 3 sets of 10 unilateral isokinetic knee extension repetitions at 60°/s. The rest intervals between sets were 1 and 2 minutes and were counterbalanced across 2 testing days, separated by a minimum of 48 hours. The work-to-rest ratio was 1:3 and 1:6. All subjects were not involved in exercise programs that included resistance exercises within the last 6 months. Statistical evaluation of the data was performed using a 2x 2 x 3 mixed factor repeated measures ANOVA [age (younger and older) x rest interval (1 and 2 min) x set (1st, 2nd, and 3rd)]. Statistical significance was set at p < 0.05 for all comparisons.

ELIGIBILITY:
Inclusion Criteria:

* Less than 75 years
* Independent

Exclusion Criteria:

* History of cardiovascular disease
* Hypertension
* Orthopedic disease

Ages: 20 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2005-02; Primary Completion 2006-03 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Peak Torque | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Martim Bottaro, PhD, Principal Investigator — University of Brasilia
Locations (1):
- University of Brasilia, Brasília, Federal District, Brazil